CLINICAL TRIAL: NCT05759169
Title: The Effect of Foot Bath Applied to Patients Receiving Hemodialysis Treatment on Comfort, Fatigue, and Dialysis Symptoms
Brief Title: The Effect of Foot Bath on Comfort, Fatigue, and Dialysis Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Sevil Şahin, Assoc Prof Dr, TC Erciyes University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021/4587
Record Dates: First submitted 2023-01-24; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Comfort; Fatigue; Symptoms and Signs
Keywords: comfort; fatigue,; foot bath; hemodialysis; nursing
MeSH Terms: conditions — Fatigue; Signs and Symptoms

STUDY DESIGN:
Intervention Model Description: This study was done in a randomized controlled experimental research pattern to determine the effect of the foot bath applied in the last 30 minutes of dialysis treatment on comfort, fatigue and dialysis symptoms for hemodialysis patients.
Masking Description: No masking done
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): In line with the literature and expert opinions, each dialysis application has been applied to individuals for 30 minutes for the first 30 minutes of 4 weeks, with a 40-43°C hot water-filled foot wash tub, placing both feet of the individual (Afrasiabifar et al., 2022; Kim et al., 2021 Shafeik et al., 2018). The researcher implemented the voluntary consent Form, Patient Demonstration Form, foot Bath Application Monitoring Chart, fatigue VAS Scale Form, dialysis Symptom Index and Hemodialysis Comfort Scale in person. At the end of the fourth week, the researcher refilled the foot Bath Application Monitoring Chart, the fatigue VAS Scale Form, the dialysis Symptom Index, and the Hemodialysis Comfort Scale. A total of 12 sessions have been performed in the foot bath, including during each dialysis treatment for 4 weeks.
  Interventions: Other: Foot Bath Tub
- Control (No Intervention): Patients in the control group have been informed about the voluntary Form, Patient Demonstration Form, fatigue VAS Scale Form, dialysis Symptom Index, and Hemodialysis Comfort Scale performed by the researcher in person. At this stage, no attempt was made to the control group at the end of the fourth week; during the last hemodialysis session, the researcher, with the fatigue VAS Scale Form, the dialysis Symptom Index and the Hemodialysis Comfort Scale face-to-face, treated the patients.

INTERVENTIONS:
Other: Foot Bath Tub — A foot bath is generally a form of rest and care where feet are put in water. Feet are body areas where fatigue is most felt as organs that carry the body's total weight. This study uses a specially designed foot bath bath bath bath to give the patients in the experimental group foot bath. The cuvette has four-stage water heating (35-45°C). It has a magnetic field and operates at 390 Watts. It has a splash guard. The sole features non-slip rubber feet. It has a heat shield feature because it has a double wall construction for heat isolation.
  Arms: Intervention

SUMMARY:
This study aimed to evaluate the effect of warm water foot baths on comfort, fatigue, and dialysis symptoms in patients undergoing hemodialysis.

This study was conducted as a randomized controlled trial. Data were collected with a total of 58 patients,31 in the intervention group and 27 in the placebo group. The data in the study is collected using the intervention and control group informed volunteer Form, Patient Demonstration Form, foot Bath Application Monitoring Chart, fatigue VAS Scale Form, dialysis Symptom Index, and Hemodialysis Comfort Scale.

DETAILED DESCRIPTION:
After obtaining the necessary permissions for the work to be performed, the researcher explained the purpose of working, and the researcher took the purpose of the work. The voluntary consent of the individuals was provided in verbal and written writing.

The researcher discussed the health team in dialysis centers to ensure that the study was carried out systematically and regularly, providing information on the purpose of the study. The forms to be applied to patients are filled by the researcher using the method of a face-to-face interview and the records obtained from the patient files.

Procedures administered to control groups:

Patients in the control group have been informed about the voluntary Form, Patient Demonstration Form, fatigue VAS Scale Form, dialysis Symptom Index, and Hemodialysis Comfort Scale performed by the researcher in person. At this stage, no attempt was made to the control group at the end of the fourth week; during the last hemodialysis session, the researcher, with the fatigue VAS Scale Form, the dialysis Symptom Index and the Hemodialysis Comfort Scale face-to-face, treated the patients.

Procedures administered to intervention groups:

In line with the literature and expert opinions, each dialysis application has been applied to individuals for 30 minutes for the first 30 minutes of 4 weeks, with a 40-43°C hot water-filled foot wash tub, placing both feet of the individual (Afrasiabifar et al., 2022; Kim et al., 2021 Shafeik et al., 2018). The researcher implemented the voluntary consent Form, Patient Demonstration Form, foot Bath Application Monitoring Chart, fatigue VAS Scale Form, dialysis Symptom Index and Hemodialysis Comfort Scale in person. At the end of the fourth week, the researcher refilled the foot Bath Application Monitoring Chart, the fatigue VAS Scale Form, the dialysis Symptom Index, and the Hemodialysis Comfort Scale. A total of 12 sessions have been performed in the foot bath, including during each dialysis treatment for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old,
* For patients over 65 years of age, the standardized Mini-mental Test (SMMT) value is 24 points or higher,
* Without pregnancy,
* With at least 6 months in HD units and 3 sessions per week,
* Continuing dialysis treatment in the same institution,
* No change in the foot bath treatment process and during the research process,
* Individuals who understand and communicate in Turkish have been investigated

Exclusion Criteria:

* Any psychiatric illness,
* Patients with neurovascular complications, advanced diabetes Mellitus,
* Patients with disease and treatment that trigger fatigue (advanced COPD, cancer, chemotherapy, and radiotherapy patients),
* With open wounds, neuropathy, etc., lower leg problems, which will prevent hot water treatment,
* Patients with peripheral vascular diseases in feet and legs,
* Also, patients with sensory deficits and foot ulcers,
* Patients using any complementary and integral treatment method during research,
* Patients with a standardized Mini-mental Test (SMMT) value of 23 points and less than 65 years old have been excluded from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Fatigue VAS Scale Form | One mounth. Fatigue levels are at the end of the process and 4 before the application begins. During the last hemodialysis session of the week, fatigue was evaluated by the VAS Scale Form.
  The rating of fatigue levels has been expressed to patients that there is no fatigue for 0 points. In comparison, 10 points indicate fatigue is very severe and are questioned how many points they have given to patients for fatigue levels.
Dialysis Symptom Index | One mounth. In the first week of the trial and 4 weeks later
  DSI contains 30 symptoms that define a specific physical or emotional symptom. Symptoms in the last seven days have been answered as yes-no, and no indicates no symptoms, and yes, that symptom has occurred. If the patient's response is yes, how much the symptom affects is evaluated by a five-type Likert scale. 1 = none, 5 = too many ratings are made. Total scale points are collected. This value varies between 0 and 150. The total scores received show an increase in the effect of the symptom mentioned as approaching 150.
Hemodialysis Comfort Scale | One mounth. In the first week of the trial and 4 weeks later
  Falcon Orak and Ark. Hemodialysis Comfort Scale (HCS), developed in 2017, with validity reliability, is a reliable scale used to assess the comfort of patients who have had hemodialysis treatment for at least six months. The hemodialysis Comfort Scale is a five-type liquid scale and consists of 9 substances and 2 sub-dimensions. T HCS can score at least 9.00 points and up to 45.00 points; 3.00 points can be achieved at least 15.00 points maximum, relax Alt-size; at least 7.00 points and up to 30.00 points can be obtained from the bottom dimension that is defeated. The increase in the value obtained indicates the level of comfort.

CONTACTS AND LOCATIONS:
Locations (1):
- Sevil Güler, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan